CLINICAL TRIAL: NCT03059316
Title: Department of Anestheia and Intensive Care Unit,Cairo University
Brief Title: Effect of Hypotensive Anesthesia on the Perfusion Index
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Hassan Saleh, department of anesthesia and intensive care unit,Cairo university, Cairo University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: N532016
Record Dates: First submitted 2017-02-07; First posted 2017-02-23 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-01

CONDITIONS: Controlled Hypotension for Nasal Surgeries
Keywords: controlled hypotension, perfusion
MeSH Terms: interventions — Nitroglycerin; Labetalol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nitroglycerin group (Active Comparator): this group will receive nitroglycerin infusion for controlled hypotension.0.5-5ug/kg/min to keep MAP 55-65mmhg then Massimo device will be attached to the patients when MAP reached the desired level
  Interventions: Combination Product: Massimo device; Drug: Nitroglycerin drug
- labetalol group (Active Comparator): this group will receive labetalol infusion fo controlled hypotension 0.4-3mg/kg/hr to keep MAP 55-65mmhg.then Massimo device will be attached to the patients when MAP reached the desired level
  Interventions: Combination Product: Massimo device; Drug: Labetalol

INTERVENTIONS:
Combination Product: Massimo device — Massimo is a newly introduced device which can measure the peripheral organ perfusion and expressed it as perfusion index(PI).
Drug: Nitroglycerin drug — Nitroglycerin is a drug used as an hypotensive agent through its vasodilation effect on veins
  Other Names: tridil
  Arms: nitroglycerin group
Drug: Labetalol — Labetalol is an antagonist of adrenergic receptors (a1, b1, b2) which is used as an hypotensive inducer. This drug targets the beta receptors 5 to 10 times more specific than alpha receptors so that minor tachycardia happens
  Other Names: trendate
  Arms: labetalol group

SUMMARY:
Controlled hypotension has been used as a mean of reducing intraoperative blood loss and better visualization of the surgical field in nasal surgeries. Perfusion index has been considered a useful tool for monitoring changes in peripheral perfusion using Masimo set and serum lactate for central perfusion. Many medications were used to induce hypotension. In this study we will compare the effects of tridil and labetalol on the perfusion.

DETAILED DESCRIPTION:
The purpose of this study to detect the degree of hypotension that helps the surgeon and dosen't impair patient's perfusion and to compare the hypotensive effects of both tridil and labetalol infusions on the perfusion.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II males and females aged 18-45 years who were scheduled for Functional Endoscopic sinus surgery (FESS)

Exclusion Criteria:

* uncontrolled hypertension, cerebrovascular disorders, bleeding and coagulation disorders, coronary artery diseases, renal or hepatic diseases or known hypersensitivity to the drugs used and pregnant.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-21 (Actual)

PRIMARY OUTCOMES:
perfusion index | 3hrs
  perfusion index is an indication of peripheral perfusion
serum lactate level | 3hrs
  lactate level is an indication of central perfusion

SECONDARY OUTCOMES:
surgical feild score | 3hrs
  isan indication of adequacy of controlled hypotension

IPD SHARING:
Plan to Share IPD: No